CLINICAL TRIAL: NCT03405948
Title: Efficiency of Botulinum Toxin Injection for Spastic Equinovarus Foot in Post Stroke Hemiparetic Patients Randomized Controlled Trial Versus Placebo
Brief Title: Efficiency of Botulinum Toxin Injection for Spastic Equinovarus Foot in Post Stroke Hemiparetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-21
Record Dates: First submitted 2017-10-31; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-10

CONDITIONS: Spastic Equinovarus Foot

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- botulinum toxin (Experimental): injection of Botulinum toxin
  Interventions: Drug: Intra muscular injection of Botulinum toxin
- placebo (Placebo Comparator): Injection of saline serum (placebo)
  Interventions: Drug: Intra muscular injection of Botulinum toxin

INTERVENTIONS:
Drug: Intra muscular injection of Botulinum toxin — posture and gait analysis were performed before injection and 4 to 6 weeks after injection

SUMMARY:
Botulinum toxin is the main treatment for focal spasticity but the effects of botulinum toxin injections with respect to limitations of gait activities are still discussed. The aim of this study is to to investigate the effects of intramuscular Botulinum toxin type A injections on quantitative gait parameters (gait speed, step length and width, single support time) and posture, in hemiparetic post stroke patients with lower limb spasticity.

DETAILED DESCRIPTION:
Multicenter, randomized, active treatment versus placebo, double-blind trial.

Hemiplegia by stroke is the leading cause of disability in adults in France (145 new cases per 100 000 population), a source of locomotor disabilities. The spastic equinovarus foot is the main cause of standing and walking disorders in these patients. Current therapies rely mainly on rehabilitation and equipment care, or for some on surgery. Botulinum toxin A is more and more used in this context. Two randomized studies (double-blind, placebo-controlled) have already demonstrated efficacy in terms of impairment (spasticity assessed using the Ashworth scale), but not in terms of capacity (evaluated from walking speed). ). The ability to maintain standing balance during an attention task and during walking, the study of quality of life have never been studied. But these parameters are important in the approach of the evaluation of such a therapy.

The purpose of the research is to evaluate the efficacy of botulinum toxin A in the treatment of adult post-stroke spastic equine varus foot in terms of: ability to maintain upright balance during an attentional task (main objective), coordination of posture and movement, standing posture, impairments and abilities, or quality of life (secondary objectives). To evaluate the tolerance and the undesirable effects related to the use of the toxin.

Methodology Prospective, comparative and randomized study, active product (botulinum toxin A) versus placebo. Patients will be recruited from the functional rehabilitation clinic. After verification of the inclusion criteria, the pre-therapeutic evaluation will be organized including: double spots, coordination posture and movement, standing posture, deficiencies and abilities, quality of life. The doctor will schedule the therapeutic session within 2 weeks. A second post-treatment evaluation will be carried out at the 4th week of follow-up according to the same scheme. The number of subjects required has been set at 84.

Method Clinical evaluation, posture and gait analysis were performed before injection and 4 to 6 weeks after injection. Quantitative gait parameters (gait speed, step length and width, single support time) were recorded with the Gaitrite walking mat. Posture was recorded with AMTI® forceplate.

Expected results: demonstrate the effectiveness of botulinum toxin on gait and balance First study about effects of botulinum toxin injection on gait parameters registered by a walking mat and objective measure of posture in dual task condition in chronic post stroke patients

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke hemiplegic patients presenting lower limb spasticity
* A minimum 12-month interval since stroke,
* Lower limb spasticity with a Modified Ashworth Scale greater than or equal to 2 on the triceps surae
* Minimum 6-month interval since a previous BTx-A injection
* To be older than 18 years.
* Patients must have an indication of treatment with Botulinum toxin, determined by a Physical and Rehabilitation Medicine specialist, based on clinical examination and gait analysis

Exclusion Criteria:

* Contraindication to the use of botulinum toxin: Myastenia, Lambert Eaton syndrome, ALS, pregnancy, breast-feeding, treatment with aminoglycoside, cyclosporine, previous hypersensitivity to botulinum toxin
* Contraindication to intramuscular injections
* Patients unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-05-19 (Actual); Primary Completion 2009-05-18 (Actual); Study Completion 2010-11-17 (Actual)

PRIMARY OUTCOMES:
Posture | 6 weeks after injection
  sway area of the center of pressure measured with AMTI® force plate

SECONDARY OUTCOMES:
Gait | 6 weeks after injection
  Walking speed measured with Gaitrite® walking mat

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Hôpital de la Timone Assistance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Kerzoncuf M, Viton JM, Pellas F, Cotinat M, Calmels P, Milhe de Bovis V, Delarque A, Bensoussan L. Poststroke Postural Sway Improved by Botulinum Toxin: A Multicenter Randomized Double-blind Controlled Trial. Arch Phys Med Rehabil. 2020 Feb;101(2):242-248. doi: 10.1016/j.apmr.2019.04.024. Epub 2019 Aug 27. PMID 31469982